CLINICAL TRIAL: NCT06741696
Title: Does Saline Irrigation At Different Temperatures Affect Pain, Edema, and Trismus After Impacted Third Molar Surgery: a Clinical Trial
Brief Title: Saline At Different Temperatures After 3rd Molar Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Armed Forces Institute of Dentistry, Pakistan (Other)
Responsible Party: Principal Investigator, Hafsa Razzaq, Dr Hafsa Razzaq, RESIDENT ORAL MAXILLOFACIAL SURGERY, Armed Forces Institute of Dentistry, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Impacted 3rd molar
Record Dates: First submitted 2024-10-24; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Post Operative Pain, Acute
Keywords: 3rd molar surgery, saline irrigation at different temperatures
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group 1 (Other): randomly selected group 1
  Interventions: Procedure: Surgical extraction; Procedure: saline irrigations
- group 2 (Other): randomly selected group 2
  Interventions: Procedure: Surgical extraction; Procedure: saline irrigations

INTERVENTIONS:
Procedure: Surgical extraction — saline irrigation at different temperatures
Procedure: saline irrigations — saline irrigation done after 3rd molar surgery

SUMMARY:
This double-blind, single-center, split-mouth, randomized prospective clinical trial was conducted among 48 systemically and periodontally healthy patients who had bilaterally asymptomatic mandibular third molars.

DETAILED DESCRIPTION:
Patients were randomly allocated into 2 groups (n = 24) according to the temperature of the saline used. In each patient, one impacted third molar was determined as the test group Trismus and swelling were evaluated on the 1st, 3rd, and 7th days postoperatively. Pain perception by visual analog scale (VAS) and the total number of analgesics taken during the 7 postoperative days were recorded. Data were analyzed using the Shapiro-Wilk test, the chi-square test, one-way analysis of variance, Duncan test, the Kruskal-Wallis test, the Dunn test, and the Friedman test (P < .05).

ELIGIBILITY:
Inclusion Criteria:1. Patients who met the requirements of the study, such as attending follow-up sessions and signing the informed consent. 2. Patients with bilateral mandibular asymptomatic vertical third molar teeth with impaction of Class I, level C.22 3. Patients who did not have any significant medical diseases or drug use, were not pregnant, had no allergy, and did not smoke.

-

Exclusion Criteria:

1 Patients with complicating systemic disease ( American Society of Anesthesiologists : 3- 6). 2. Patients who have second molars with severe periodontal defect or deep periodontal pocket (probing depth >4 mm). 3. Patients with poor oral hygiene. 4. Patients with a history of using analgesics 12 hours ago or antibiotics 1 month before. 5. The presence of cysts or tumors around the impacted third molar.

-

Max Age: 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
post operative pain after 3rd molar surgery | 7 days
  Trismus and swelling were evaluated on the 1st, 3rd, and 7th days postoperatively. Pain perception by visual analog scale (VAS) and the total number of analgesics taken during the 7 postoperative days were recorded

CONTACTS AND LOCATIONS:
Overall Officials: hafsa razzaq razzaq, BDS, Principal Investigator — Armed Forces Institute of Dentistry , Rawalpindi
Locations (1):
- Armed Forces Institute of Dentistry, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No